CLINICAL TRIAL: NCT06321107
Title: A Phase II/III Extension Study Comparing the Long-term Safety of GenSci094 and Gonal-f® in Chinese ART Patients
Brief Title: Long-term Follow-up Safety of a Single Injection of GenSci094 for Ovarian Stimulation Using Daily Recombinant FSH as Reference
Status: Active, not recruiting | Type: Observational
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: GenSci094-304
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group: Gensci094
- Control group: rFSH

SUMMARY:
The purpose of this study is to evaluate the safety of a single injection of GenSci094 during Controlled Ovarian Stimulation up to 1 year old of the infants from previous studies.

DETAILED DESCRIPTION:
Two previous RCTs (a phase II and phase III studies of GenSci094, one is NCT06091436) investigated if a single injection of GenSci094 was non-inferior to daily treatment with recFSH in initiating multi-follicular growth. The two studies followed 12 weeks after embryo transfer. This study is a follow-up to the above mentioned RCTs. The purpose of this study is to follow-up with participants of the original study to determine the long-term effect a single injection of GenSci094 during Controlled Ovarian Stimulation might have on newborns until they are 1 year old.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign informed consent
2. Subjects who participated in Phase II or Phase III clinical trial of GenSci094 and received at least one treatment with GenSci094 or Gonal-F ®
3. Subjects who indentified an ongoing pregnancy in Phase II or Phase III clinical trial of GenSci094

Exclusion Criteria:

NA

Ages: 20 Years to 39 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Subjects who indentified an ongoing pregnancy in Phase II or Phase III clinical trial of GenSci094
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Summary of Pregnancy Outcome | To be assessed at late abortion or birth (up to 10 months)
  Pregnancy outcomes were reported at the optional long-term follow up visit.

SECONDARY OUTCOMES:
neonatal birth outcomes | To be assessed at birth (up to 10 months)
  To be assessed by the birth attendant/ Obgyne
Infant development | up to infant age 12 months
  To assess infant's development, weight in grams/kilograms, height in centimeters and head circumference in centimeters are measured.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Liang, doctor, Study Chair — The Sixth Affiliated Hospital, Sun Yat-sen University Guangdong Gastrointestinal Hospital
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University Guangdong Gastrointestinal Hospital, Guangzhou, Guangdong, China